CLINICAL TRIAL: NCT01696487
Title: Impact of Fructose Consumption on Intestinal Permeability in Non-alcoholic Fatty Liver Disease (NAFLD) - a Pilot Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: State Government of Vienna, Austria (Medizinisch-Wissenschaftlicher Fonds des Bürgermeisters der Bundeshauptstadt Wien) (Unknown)
Responsible Party: Principal Investigator, Prof. Michael Trauner, MD, Professor, MD, Head and Chair of the Division of Gastroenterology and Hepatology, Department of Internal Medicine III, Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Fru1.0
Record Dates: First submitted 2012-09-01; First posted 2012-10-01 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Non-alcoholic Fatty Liver Disease; Non-alcoholic Steatohepatitis
Keywords: non-alcoholic fatty liver disease; non-alcoholic steatohepatitis; NAFLD; NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Healthy Volunteers (Experimental): Volunteers will be challenged with oral 150g Fructose per day for 28 days.
  Interventions: Dietary Supplement: High oral Fructose challenge (150g per day for 28 days)
- NAFLD (No Intervention): Patients with confirmed fatty liver (imaging positive) will be compared at baseline with other arms.
- NASH (No Intervention): Patients with confirmed non-alcoholic steatohepatitis (biopsy proven) will be compared at baseline with other arms.
- Hepatitis C genotype 1 (HCV-GT1) (No Intervention): Patients with confirmed hepatitis C genotype 1 will be compared at baseline with other arms and act as different liver disease control group

INTERVENTIONS:
Dietary Supplement: High oral Fructose challenge (150g per day for 28 days)
  Arms: Healthy Volunteers

SUMMARY:
The spectrum of NAFLD as emerging epidemic ranges from steatosis to steatohepatitis (NASH), cirrhosis and hepatocellular carcinoma (HCC). Disease progression is poorly understood and treatment options are limited. Fructose overconsumption has been associated with gut permeability and progression of NAFLD. To unravel the mechanisms of fructose-induced intestinal changes, volunteers will receive a 4-week fructose challenge prior to assessment of intestinal permeability/translocation using endomicroscopy, sugar probes, serum markers of intestinal damage, inflammation, iron/copper homeostasis and histological/molecular analysis of intestinal biopsies. Findings in volunteers will be compared with liver patients undergoing study procedures without fructose challenge. Translational in vitro experiments will explore cellular responses to fructose and endotoxin. This project should provide novel insights into dietary induced alterations of the gut integrity in progression of NAFLD to NASH.

ELIGIBILITY:
1. Healthy men and women from 18 to 85, no disease history, no intake of regular medication.
2. Patients with confirmed (at least one imaging positive) intrahepatic fat accumulation (NAFL), male and female
3. Patients with confirmed NASH (biopsy within 6 months prior to study), male and female
4. Diagnosed HCV, genotype 1, male and female

Signed informed consent

General exclusion criteria (for all groups)

1. Pregnancy and lactation
2. Imprisoned persons
3. Inflammatory bowel conditions (celiac disease, Crohn's disease, ulcerative colitis)
4. Prior bariatric surgery
5. Alcoholic steatohepatitis and/or alcohol consumption > 140 gramms per week (or > 30g/day)
6. Other liver diseases (autoimmune, genetic, cholestatic, Wilson disease, Weber-Christian disease, partial lipodystrophy of the face sparing type, abetalipoproteinemia, and jejunal diverticulosis with bacterial overgrowth.)
7. Virus hepatitis (A, B, C) (except for group (4): defined as HCV, genotype 1)
8. Known allergic reaction to the drugs used (see material and methods)
9. Intake of drugs known to accumulate intrahepatic lipids (e.g. steroids/glucocorticoids, tamoxifen, amiodarone, perhexiline maleate, synthetic estrogens, antiretroviral agents, tetracycline, minocycline, certain pesticides, methotrexate)
10. Intake of drugs known to drive fibrosis/cirrhosis (e.g. azathioprine, oral contraceptive pills)
11. Inability or contraindications to perform study procedures
12. General and absolute endoscopy contraindications

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Gaps per 1000 intestinal epithelial cells assessed by confocal laser endomicroscopy | Time point 1 (day 1 - all study groups)
  Gaps per 1000 intestinal cells will be assesed during gastroscopy by confocal laser endomicroscopy at time point 1 in all study groups and after the 4 week fructose challange in healthy volunteers only
Gaps per 1000 intestinal epithelial cells assessed by confocal laser endomicroscopy | point 2 (week4/day28 - after fructose challange; healthy volunteers only)
  Gaps per 1000 intestinal cells will be assesed during gastroscopy by confocal laser endomicroscopy at time point 1 in all study groups and after the 4 week fructose challange in healthy volunteers only

CONTACTS AND LOCATIONS:
Overall Officials: Michael Trauner, MD, Principal Investigator — Division of Gastroenterology and Hepatology Department of Internal Medicine III Medical University of Vienna
Locations (1):
- Medical University of Vienna, General Hospital of Vienna, Vienna, Austria